CLINICAL TRIAL: NCT05629754
Title: Long-term Outcomes and Development of Retropatellar Chondropathy After Tibial Tubercle Distomedialisation for Patellar Maltracking and Patella Alta Without Instability: 10 Year Follow-up of a Prospective Cohort
Brief Title: 10-year Follow-up After Tibial Tubercle Transposition
Acronym: TTTfollow-up
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre for Orthopaedic Research Alkmaar (Other)
Collaborators: Noordwest Ziekenhuisgroep (Other)
Responsible Party: Principal Investigator, Joyce L Benner, PhD, Principal Investigator, Centre for Orthopaedic Research Alkmaar
Other Study IDs: NL82613.029.22
Record Dates: First submitted 2022-11-09; First posted 2022-11-29 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Tibial tubercle transfer; Long-term follow-up
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI, radiological assessment — MRI and radiological assessment of the involved knee

SUMMARY:
Patellofemoral pain is a common complaint especially in young adults. It can be caused by patellar maltracking. Part of this is a patella alta. When patellar maltracking is the cause of the problem and conservative therapy fails, surgery, a tibial tuberosity transposition, may be considered. Most research has been done in patients with recurrent patella luxation. However, in patients without luxation, research is scarce.

It is known that patients with patella alta have an increased risk of developing patellofemoral chondropathy due to increased pressure. With this study, we aim to investigate whether and how a tibial tuberosity transposition in patients with patella alta and no instability affects the degree of patellofemoral chondropathy and patient satisfaction after 10 years. This will allow us to educate patients regarding long-term outcomes better.

DETAILED DESCRIPTION:
Anterior knee pain is a common complaint, especially in younger and active adults. An obvious source for anterior knee pain is patellar maltracking, which is often associated with patella alta (a high-riding patella). Due to maltracking, the cartilage of the patella can face a greater amount of pressure, which can cause cartilage damage. When conservative treatment fails, a surgical intervention can be considered. One of the surgical options is performing a tibial tubercle transfer (TTT), where the patella is being distalized and medialized. As a result, the improvement in patellar tracking will reduce the pressure on the retropatellar cartilage. The TTT has been proven effective in patients with patellar instability but less is known about patients without instability. Specifically, whether these patients face a higher risk of developing retropatellar cartilage damage ('retropatellar chondropathy') due to this intervention is currently unknown.

The primary aim of this study is to determine the incidence and the degree of retropatellar chondropathy 10 years after a TTT in patients with anterior knee pain without patellar instability. The secondary aim is to evaluate the long-term patient reported outcomes (PROMs) 10 years after a TTT in patients with anterior knee pain without patellar instability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Participated in an earlier cohort study
* Underwent a tibial tubercle transposition between 2012 and 2015
* Preoperative MRI available

Exclusion Criteria:

* No preoperative MRI is available
* Patellar-related surgery after the initial surgery
* Female patients that are (expecting to be) pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whom around 10 years ago presented with anterior knee pain and patella maltracking without instability, where conservative therapy failed and a TTT was performed, and who participated in the original cohort.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-11-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Modified Outerbridge Classification | 10-year follow-up assessment
  Degree of retropatellar cartilage damage

SECONDARY OUTCOMES:
Patellar height | 10-year follow-up assessment
  Patellar height measured by radiological assessment lateral view
Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire | 10-year follow-up assessment
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Kujala Anterior Knee Pain Score (AKPS) questionnaire | One measurement
  The Kujala AKPS is a 13-item screening instrument designed to assess patellofemoral pain in adolescents and young adults, with a variable ordinal response format (e.g., no pain (5) to constant pain (0)). Total scores range from 0 to 100, with a higher score indicating less symptoms.
Visual Analogue Scale (VAS) for pain | 10-year follow-up assessment
  The pain VAS is a unidimensional measure of pain intensity, scored from 0 (no pain) to 100 (highest possible pain intensity).

CONTACTS AND LOCATIONS:
Overall Officials: JL Benner, PhD, Principal Investigator — Noordwest Ziekenhuisgroep
Locations (1):
- Noordwest Ziekenhuisgroep, Alkmaar, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bayoumi T, van Duijvenbode DC, Benner JL, Boerma-Argelo KDS, Stavenuiter MHJ, van der List JP. Clinical Improvement Is Achieved Following Tibial Tubercle Distomedialization for Patellar Maltracking and Patella Alta Without Instability. Arthrosc Sports Med Rehabil. 2021 Jun 15;3(3):e845-e853. doi: 10.1016/j.asmr.2021.01.027. eCollection 2021 Jun. PMID 34195653